CLINICAL TRIAL: NCT01221077
Title: A Randomized, Double-Blind, Phase 2 Study of Erlotinib (Tarceva®) in Combination With OSI-906 or Placebo in Chemonaive Patients With Advanced NSCLC With Activating Mutations of the Epidermal Growth Factor Receptor (EGFR) Gene
Brief Title: Study of Erlotinib (Tarceva®) in Combination With OSI-906 in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) With Activating Mutations of the Epidermal Growth Factor Receptor (EGFR) Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSI-906-207
Record Dates: First submitted 2010-10-05; First posted 2010-10-14 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; Non Small Cell Lung Cancer
Keywords: NSCLC; Epidermal Growth Factor Receptor; EGFR; Non-small cell lung cancer; Tarceva; Activating mutations; OSI-906; Chemonaive; IGF-IR; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Erlotinib plus OSI-906 (Experimental): As of 01 March 2013, OSI-906 is no longer being administered
  Interventions: Drug: OSI-906; Drug: Erlotinib
- Arm B: Erlotinib plus Placebo (Placebo Comparator): As of 01 March 2013, the matching placebo is no longer being administered
  Interventions: Drug: Erlotinib; Drug: Placebo

INTERVENTIONS:
Drug: OSI-906 — As of 01 March 2013, OSI-906 is no longer being administered
  Arms: Arm A: Erlotinib plus OSI-906
Drug: Erlotinib — Erlotinib administered orally
  Other Names: OSI-774; Tarceva
Drug: Placebo — As of 01 March 2013, the matching placebo is no longer being administered
  Arms: Arm B: Erlotinib plus Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase 2 study of Erlotinib (Tarceva®) in combination with OSI-906 in Patients with Advanced non-small cell lung cancer (NSCLC) with Activating Mutations of the Epidermal Growth Factor Receptor (EGFR) Gene who are Chemonaive.

DETAILED DESCRIPTION:
Based on the recommendation of the Data Monitoring Committee, OSI-906 and matching placebo are no longer being administered as of 01 March 2013.

This is a multi-center, randomized (1:1), double-blind, placebo-controlled, phase 2 study. Patients will be stratified according to the following 2 parameters: (1) EGFR activating mutation type (exon 19 deletion versus exon 21 single point mutation); and (2) Eastern Cooperative Oncology Group (ECOG) performance status (0 vs. 1).

ELIGIBILITY:
Inclusion Criteria:

* Historically confirmed advanced NSCLC stages IIIB or IV
* Exon 19 deletion or exon 21 activating mutation in EGFR
* EGFR mutation status must be confirmed for participation in the study. EGFR can be performed either by central or local laboratory. If analysis is done locally, verifiable documentation confirming the EGFR mutation status must be submitted for review and approval by sponsor prior to randomization. If no local result is available, formalin-fixed, paraffin-embedded archival tissue representative of the tumor or, in the absence of archival tissue, a fresh tumor tissue sample of sufficient size to perform EGFR mutation analysis must be submitted centrally. Results of the central analysis must be available prior to randomization. Additionally, subjects should provide tissue blocks for biomarker central analysis whenever possible. Ideal tissue requirement: block with ≥5 mm2 tumor area sufficient to provide four 4-micron, and five 10-micron sections
* Measurable disease according to RECIST (version 1.1)
* ECOG performance status 0-1
* Must be able to take oral medication
* Fasting glucose <= 150 mg/dL (8.3 mmol/L). Concurrent use of non-insulinotropic anti hyperglycemic therapy is permitted if the dose has been stable for >= 4 weeks at the time of randomization
* Adequate hematopoietic, hepatic, and renal function as follows:

  * Neutrophil count >= 1500/uL
  * Platelet count >= 100,000/uL
  * Serum creatinine <= 1.5 x Upper Limit of Normal (ULN)
  * Potassium, magnesium, and calcium within normal limits (supplementation and re-testing is permitted)
  * Total bilirubin <= 1.5 x ULN
  * AST and ALT <= 2.5 x ULN, or <= 5 x ULN if patient has documented liver metastases
* Female subject must be either:

  * Of non child bearing potential:

    1. post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
    2. documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening).
  * Or, if of childbearing potential:

    1. must have a negative urine pregnancy test at Screening, and
    2. must use two forms of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 30 days after final study drug administration. Acceptable forms include:

       1. Established use of oral, injected or implanted hormonal methods of contraception;
       2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
       3. Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Female subject must not be breastfeeding at Screening or during the study period and for 30 days after final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period and for 30 days after final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 30 days after final study drug administration. Acceptable forms include:

  1. Established use of oral, injected or implanted hormonal methods of contraception.
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  3. Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Male subjects must not donate sperm starting at Screening and throughout the study period and for at least 30 days after final study drug administration.
* Patients must provide written informed consent to participate in the study
* Patients may not have received chemotherapy for advanced NSCLC. Previous adjuvant and/or neoadjuvant treatment for NSCLC is permitted
* Prior radiation therapy is permitted provided patients have recovered from the acute, toxic effects of radiotherapy prior to randomization. A minimum of 28 days must have elapsed between the end of radiotherapy and randomization
* Prior surgery is permitted provided that the surgery was done >= 28 days prior to randomization and adequate wound healing has occurred prior to randomization

Exclusion Criteria:

* Prior exposure to agents directed at the Human Epidermal Receptor (HER) axis (eg, erlotinib, gefitinib, and cetuximab)
* Prior insulin-like growth factor -1 receptor (IGF-1R) inhibitor therapy
* Malignancies other than NSCLC within the past 3 years (exceptions if curatively treated; basal or squamous cell carcinoma of skin; locally advanced prostate cancer; ductal carcinoma in situ of breast; in situ cervical carcinoma; and superficial bladder cancer)
* Diabetes mellitus currently requiring insulinotropic or insulin therapy
* Use of proton pump inhibitors such as omeprazole within 14 days prior to randomization. H2-receptor antagonists such as ranitidine are not excluded
* Symptomatic brain metastases that are not stable, require steroids, or have required radiation and/or other related treatment (i.e., anti-epileptic medication) within 21 days prior to randomization
* Participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives whichever is longer, prior to the initiation of Screening or during the course of the study.
* History of poorly controlled gastrointestinal disorders that could affect the absorption of study drug (eg, Crohn's disease or ulcerative colitis)
* History (within last 6 months) of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac disease includes second/third degree heart block; clinically significant ischemic heart disease; superior vena cava (SVC) syndrome; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but no ordinary physical activity results in fatigue, palpitation, or dyspnea)
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (>= grade 3), left bundle branch block (LBBB), or asymptomatic sustained ventricular tachycardia are not allowed. Patients with atrial fibrillation controlled by medication are not excluded
* Mean QTcF interval >= 450 msec at screening
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) ('Torsades List' on www.azcert.org/medical-pros/drug-lists/bycategory.cfm) are prohibited within 14 days prior to randomization
* Use of strong/moderate CYP1A2 inhibitors such as ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded
* Use of strong/moderate CYP3A4 inhibitors and inducers
* History of cerebrovascular accident (CVA) within 6 months prior to randomization or that resulted in ongoing neurologic instability
* History of any psychiatric or neurologic condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug
* Active infection, serious underlying medical condition (including any type of active seizure disorder within 12 months prior to randomization), symptomatic brain metastases, or serious chronic illness that would impair the ability of the patient to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-04-08 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of OSI-906 in combination with Erlotinib or Erlotinib plus placebo | 15 months
  Time from randomization to disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by investigator or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 33 months
  Time from the date of randomization until the documented date of death.
Disease Control Rate (DCR) | 33 months
  Proportion of patients with a best overall response of complete response (CR), partial response (PR), or stable disease based on RECIST version 1.1 criteria.
Best Overall Response Rate | 33 months
Duration of Response (CR/PR) | 33 months
  Time from the date of the first documented response (CR/PR) to documented progression or death due to underlying cancer.
  Defined for patients whose best overall response was CR or PR.
Safety assessed through evaluation of adverse events, laboratory, physical examination, and Electrocardiogram (ECG) data | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (29):
- United States (13):
  - University of California, San Diego/Moores Cancer Center, La Jolla, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance University of Washington, Seattle, Washington
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Singapore (2):
  - Oncocare Cancer Center, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Ilsimri, Hwasun-gun
  - Asan Medical Center, Songpa-gu, Seoul
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
- Thailand (4):
  - National Cancer Institute, Phayathai, Bangkok
  - Maharaj Nakorn Chiangmai, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Songklanagarind Hospital, Prince of Songkla University, Songkhla

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=264